CLINICAL TRIAL: NCT05659784
Title: Virtually Assisted Home Rehabilitation After Acute STroke (VAST-rehab)
Acronym: VAST-rehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Sean Savitz, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-20-0384
Record Dates: First submitted 2022-12-12; First posted 2022-12-21 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Stroke
Keywords: rehabilitation
MeSH Terms: conditions — Stroke | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telerehabilitation (Experimental)
  Interventions: Other: Telerehabilitation

INTERVENTIONS:
Other: Telerehabilitation — Education based telerehab with rehabilitation therapists providing education on home exercises and stroke specific information

SUMMARY:
The purpose of this study is to investigate the feasibility of a virtual education and virtual visit program in engaging patients with rehabilitation at home after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent provided by the subject or legally authorized representative.
* Occurrence of a hemorrhagic or ischemic stroke
* pre-stroke mRS less than 3
* Qualifying Stroke Event must be confirmed by CT or MRI
* Recommended to participate in self-guided or in-person rehabilitation activities by a physician or rehabilitation therapist
* Must have sufficient cognitive and language abilities to comprehend verbal commands and to carry out the study assessments
* Able to access the internet via a personal device

Exclusion Criteria:

* . History of neurological or other disease resulting in significant functional impairment (e.g.Parkinson's disease, motor neuron disease, moderate dementia, arthritis,contractures or fixed anatomical abnormality).
* Subjects with a severe comorbid disorder that has reasonable likelihood of limiting survival to less than 6 months.
* Any other conditions that, in the opinion of the investigators, would preclude safe and/or effective participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Feasibility as assessed by number of participants that completed all scheduled visits. | end of study(12 weeks form baseline)

SECONDARY OUTCOMES:
Change in Functional independence as assessed by the Functional Independence Measure (FIM) | Baseline, end of study (about 13-14 weeks after baseline)
  This is an 18 item questionnaire and each is scored from 1(complete dependence on helper) to 7(complete independence), a higher number indicating more independence
Patient-Specific Functional Scale | Baseline, end of study (about 13-14 weeks after baseline)
  This tool allows for Subjects to self report activities of daily living that have been affected by stroke and rate severity of impact on these activities. This is scored from 0(unable to perform activity) to 10(able to perform activity at the same level as before injury or problem)
Change in impact of stroke as assessed by the Stroke Impact Scale (SIS) | Baseline, end of study (about 13-14 weeks after baseline)
  This is a A 59 item questionnaire whereby subjects identify the impact of stroke on strength, hand function, mobility, activities of daily living, memory, communication, emotion, and handicap. Item responses are scored on a 5-point Likert-style scale. A score of 1 = an inability to complete the item and a score of 5 = no difficulty experienced at all. A standardized score ranging from 0 to 100 is calculated for all domains, with higher scores indicating a higher quality of life
Change in quality of life as assessed by the EuroQol-5-5level scale (EQ-5D-5L) | Baseline, end of study (about 13-14 weeks after baseline)
  A self reporting, quality of life measurement that asks Subjects to rate their severity of problems related to mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. There are 5 questions in the first section and each question is scored from 0-5,a higher number indicating a worse outcome .There is a visual scale at the end that is scored from 0(worst health) to 100(best health), higher number indicating better outcome .
  .
Change in cognitive impairment as assessed by the Short Montreal Cognitive Assessment(s-MoCA) | Baseline, end of study (about 13-14 weeks after baseline)
  8 item questionnaire ,with a possible score of 1-5, a lower number indicating higher cognitive impairment
Change in performance in activities of daily living as assessed by the Barthel Index | Baseline, end of study (about 13-14 weeks after baseline)
  This is a scoring technique that measures performance in ten activities of daily living including feeding, wheelchair to bed transfers, grooming ,chair to toilet transfers, walking, using stairs, dressing, and continence of bowels and bladder. This is a 10 item questionnaire and is scored from 0-100, a higher score indicating higher level of independence.
Change in symptoms related to stroke as assessed by the National Institute of Health Stroke Scale(NIHSS) | Baseline, end of study (about 13-14 weeks after baseline)
  the score for each ability is a number between 0(normal functioning) to 4(completely impaired). The score is calculated by adding the number for each element of the scale with a highest score of 42, a higher score meaning more impairment.
Change in degree of disability or dependence as measured by the Modified Rankin Score(mRS) | Baseline, end of study (about 13-14 weeks after baseline)
  mRS is a 6 point disability scale with possible scores from 0(no disability) to 5(disability requiring constant care) a higher score indicating more disability

CONTACTS AND LOCATIONS:
Overall Officials: Sean Savitz, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stevens EA, Muraly N, Da Silva CP, Richards L, Sosa A, Smith H, Richard AS, Manji S, Russell ME, Savitz SI. Virtually assisted home rehabilitation after acute stroke (VAST-rehab): A descriptive pilot study for young and underserved stroke survivors. Digit Health. 2025 Mar 17;11:20552076251324443. doi: 10.1177/20552076251324443. eCollection 2025 Jan-Dec. PMID 40103648